CLINICAL TRIAL: NCT04000204
Title: The Comparison of Safety and Effectiveness Between HYAJOINT Plus and Bioventus Durolane for the Treatment of Knee Osteoarthritis Pain
Brief Title: The Comparison of Two Crosslinked Hyaluronate for the Treatment of Osteoarthritis Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDCT-CKHP
Record Dates: First submitted 2019-06-18; First posted 2019-06-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; synovial fluid supplement; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYAJOINT Plus (Experimental)
  Interventions: Device: HYAJOINT Plus
- Durolane (Active Comparator)
  Interventions: Device: Durolane

INTERVENTIONS:
Device: HYAJOINT Plus — 60 mg / 3 ml cross-linked hyaluronan, SciVision Biotech Inc.
  Arms: HYAJOINT Plus
Device: Durolane — 60 mg / 3 ml cross-linked hyaluronan, Bioventus LLC.
  Arms: Durolane

SUMMARY:
The aim of this study is to compare the safety and effectiveness between two BDDE-crosslinked hyaluronate, HYAJOINT Plus and Durolane, for the Treatment of Knee Osteoarthritis Pain.

ELIGIBILITY:
Inclusion Criteria:

1. age from 35 to 85 years;
2. radiographic Kellgren-Lawrence grade II to III;
3. symptoms ≧6 months despite conservative treatments such as analgesics, NSAID and/or physical therapy;
4. average knee pain score ≧30mm on 100-mm visual analog scale (VAS) in recent one week;
5. radiographic evidence of bilateral knee OA not reason for exclusion if VAS pain in contralateral knee <30mm.

Exclusion Criteria:

1. previous orthopedic surgery in the lower extremity;
2. disabling osteoarthritis of hip or ankle;
3. previous IAHA within 6 months;
4. IA steroid or joint puncture within 3 months;
5. characters of severe acute synovitis under ultrasound (US) examination, such as Grade 3 in suprapatellar synovitis (SPS), suprapatellar effusion (SPE), medial compartment synovitis (MCS) or lateral compartment synovitis (LCS);
6. Any specific medical condition, such as rheumatoid arthritis, Lupus erythematous, hemiparesis, infection, neoplasm, and etc., that would interfere with assessments;
7. confirmed or suspected pregnancy or lactating;
8. known allergy history to any avian protein or HA product.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
The change from baseline VAS pain score at 6 months post-injection. | 6 months post-injection
  The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'

SECONDARY OUTCOMES:
Visual analog scale (VAS) score for pain change | Baseline, 1, 3, 9 and 12 months post-injection
  The change from baseline VAS pain score at 1, 3, 9 and 12 months post-injection. The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'
Adverse events reported from the baseline and during the study period | 1, 3, 6, 9 and 12 months post-injection
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Likert scale score change | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline WOMAC score at 1, 3, 6, 9 and 12 months post-injection. A 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Total score is 96 and lower scores indicate better outcomes.
Visual analog scale (VAS) score for stiffness change | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline VAS stiffness score at 1, 3, 6, 9 and 12 months post-injection. The VAS scale uses a 100 mm line labelled at '0' with 'no stiffness' and '100' with 'worst stiffness'.
Visual analog scale (VAS) score for satisfaction change | 1, 3, 6, 9 and 12 months post-injection
  The change from baseline VAS satisfaction score at 1, 3, 6, 9 and 12 months post-injection. Patients rate their treatment satisfaction based on a 100 mm VAS. The VAS scale uses a 100 mm line labelled at '0' with 'least satisfaction' and '100' with 'highest satisfaction'.
Timed Up-and-Go test (TUG) change | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline TUG time at 1, 3, 6, 9 and 12 months post-injection. A simple measurement of time in seconds for a subject to rise from an armchair, walk 3 meters, turn around, walk back to the chair, and sit down.
Single-leg stance test (SLS) change | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline SLS time at 1, 3, 6, 9 and 12 months post-injection. A simple measurement of time in seconds for a subject raising one foot up without touching it to the supported lower extremity with knee OA and maintain balance for as long as possible.
Knee joint inflammatory state change by ultrasonic inspection | Baseline, 1, 3, 6, 9 and 12 months post-injection
  The change from baseline of the subject knee inflammatory state at 1, 3, 6, 9 and 12 months post-injection through ultrasonic inspection.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan